CLINICAL TRIAL: NCT05320757
Title: Effects of PARP Inhibitor on Tumor Microenvironment in High-risk Endometrial Cancer Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Ka-Yu Tse, Principal Investigator, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UW 21-521
Record Dates: First submitted 2022-02-23; First posted 2022-04-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Endometrial Cancer
Keywords: Endometrial cancer, olaparib
MeSH Terms: conditions — Endometrial Neoplasms | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Olaparib (Experimental): Olaparib: 300mg BID orally for 10 - 28 days (stop 3 - 4 days before definitive treatment)
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib — a PARP inhibitor
  Other Names: Lynparza

SUMMARY:
This is a window study where treatment-naïve patients will receive olaparib before definitive treatment. The aim is to evaluate the DNA damage and inflammatory response after PARP inhibitor.

DETAILED DESCRIPTION:
Patients with high-risk endometrial cancers are prone to develop recurrence. The response rate to conventional chemotherapy in persistent or recurrent endometrial cancer is poor. Recent research demonstrated that immune checkpoint with or without targeted therapy was an effective treatment option. However, the change of immune landscape in the blood and tumor after PARPi is not clear.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be capable of giving signed informed consent
2. Patients must be at least 18 years old
3. Patients must have newly diagnosed and histologically confirmed high-risk endometrial cancer, including:

   1. G3 endometrioid, any stage
   2. Type 2 (such as serous, clear cell, carcinosarcoma), any stage
   3. G1 endometrioid, stage 2 or beyond
4. The endometrial cancer should be visible on pre-treatment ultrasound, or endometrial lining should be 5mm or above
5. An archived FFFE sample of endometrial biopsy or at least 8 unstained slides should be available
6. Patients should have Eastern Cooperative Oncology Group (ECOG) performance score 0 to 1
7. Patients must have adequate bone marrow, renal, hepatic, thyroid and neurological function within 28 days prior to administration of study treatment
8. Patients must be able to swallow oral medication
9. Patients must have a life expectancy of ≥ 16 weeks
10. Patients must either be postmenopausal or show evidence of non-childbearing status for women of childbearing potential

Exclusion Criteria:

1. Patients with other malignancy unless curatively treated with no evidence of disease for >= 5 years, are excluded.
2. Patients whose resting ECG indicating uncontrolled, potentially reversible cardiac conditions, or patients with congenital long QT syndrome, are excluded.
3. Patients with myelodysplastic syndrome/acute myeloid leukaemia or with features suggestive of MDS/AML, other hematological diseases such as venous or arterial thrombosis and thrombocytopenia are excluded.
4. Patients with symptomatic uncontrolled brain metastases are excluded.
5. Patients who are unable to swallow orally administered medication and gastrointestinal disorders are excluded.
6. Patients with immunocompromised condition, active hepatitis, or persistent toxicities caused by previous cancer therapy, are excluded.

9. Concomitant use of known strong CYP3A inhibitors or inducer are excluded. 10. Patients who have major surgery within 2 weeks, previous allogenic bone marrow transplant, are excluded.

11. Patients with a known hypersensitivity to olaparib or any of the excipients of the product are excluded.

12. Use of an investigational drug within 30 days or 5 half-lives, whichever is longer, proceeding the first dose of study drug is not allowed.

13. Pregnant or breastfeeding women are excluded. 14. Patients who are judged by the investigator to be unlikely to comply with study procedures, restrictions and requirements are excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Extent of DNA damage | Up to 18 months
  change of gH2Ax expression in tumor tissues in high-risk EC patients before and after olaparib as assessed by immunofluorescent staining (% change)

SECONDARY OUTCOMES:
Change of CD4 and CD8 T cells in tumor | Up to 18 months
  Change of T cell population in tumours before and after olaparib as assessed by immunostaining (% change)
Change of interferon gamma level in blood | Up to 18 months
  Change of interferon gamma in blood before and after olaparib as assessed by ELISA (% change)

CONTACTS AND LOCATIONS:
Overall Officials: Ka Yu Tse, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No